CLINICAL TRIAL: NCT00703508
Title: Pharmacogenetics of Metformin Action in PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM11153; 2U54HD034449 (NIH)
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Experimental): Metformin tablet, 500 mg/tablet, 2 tablets every twelve hours, 9 months duration
  Interventions: Drug: Metformin 500 mg tablet

INTERVENTIONS:
Drug: Metformin 500 mg tablet — Metformin 500 mg tablets; two tablets every 12 hours for 9 months
  Other Names: Glucophage

SUMMARY:
1. The polycystic ovary syndrome is the major cause of infertility in the United States. Metformin has been shown to increase frequency of ovulations in PCOS, and is used in clinical practice to treat infertility, but some women with PCOS do not respond to metformin treatment.
2. Knowing that a specific gene predicts the effect of metformin on ovulation would facilitate more efficient and effective treatment of infertility in PCOS.

DETAILED DESCRIPTION:
The polycystic ovary syndrome (PCOS) affects approximately 6-10% of women of childbearing age, i.e., 3.5-5.5 million women in the United States. PCOS is the most common endocrine disturbance of young women and the major cause (75%) of anovulatory infertility in the United States. We hypothesize that women with the polycystic ovary syndrome (PCOS) who have the G/G genotype of single nucleotide polymorphism (SNP)_ rs8111699 in STK11 will exhibit a significantly greater response to metformin, in terms of ovulation, compared with women with either the C/G or C/C genotype. Specifically, we anticipate the frequency of ovulation (defined by number of ovulations/9 months/subject) to be at least 2-fold higher in women with the G/G STK11 genotype compared with women with either the C/G or C/C genotype.

To test this hypothesis, we will obtain DNA for STK11 genotyping in 36 women with PCOS who are treated with metformin and carefully monitored for ovulation for 9 months. STK11 genotype status will be determined, and the ovulation rates in the G/G, G/C and C/C genotype groups will be compared with one another. Our goal is to identify the genes that predict or modify response to commonly prescribed medications that will allow physicians to better choose among existing therapies and individualize treatment. While metformin has been shown to increase ovulatory frequency in PCOS and is widely used in clinical practice to treat infertility, a substantial number of women either do not respond or are slow to respond to metformin treatment.

Knowing that a specific STK11 genotype predicts the effect of metformin on ovulation would facilitate more efficient and effective treatment of infertility in PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women between 18-45 years of age and BMI less than 42
* Diagnosed with PCOS as defined by the Rotterdam criteria, which is a combination of any two of the following three criteria: 1) chronic oligo- or amenorrhea (<8 menstrual periods annually); 2) biochemical or clinical androgen excess; and 3) polycystic ovaries on ultrasonography -Normal thyroid function tests and serum prolactin; and exclusion of 21 alpha hydroxylase deficiency by a fasting 17 alpha hydroxyprogesterone less than 200 ng/dl -In acceptable health on the basis of interview, medical history, physical examination, and laboratory tests (CBC, SMA20,urinanalysis) -Able to provide signed, witnessed informed consent -Able to comply with study requirements

Exclusion Criteria:

-Diabetes mellitus by fasting glucose or OGTT, or clinically significant pulmonary, cardiac,renal,hepatic,neurologic,psychiatric,infectious,neoplastic and malignant disease (other than non-melanoma skin cancer) -Current use of oral contraceptives; use of fertility drugs within 6 months of study -Current or recent use (within 3 months prior to study entry) of metformin -Documented or suspected recent (within one year)history of drug abuse or alcoholism -Ingestion of any investigational drug within two months prior to study onset.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2008-07; Primary Completion 2013-09 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E. Nestler, M.D., Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - University Of Virginia General Clinical Research Center, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Result] Cheang KI, Bhavi Modi, Maria Shulleeta, William S. Evans, Lubna Pal, Jerome F. Strauss and John E. Nestler: Genetic Polymorphisms and Ovulatory Responsiveness to Metformin in Women with Polycystic Ovary Syndrome. Endo Reviews 36 (2): Supplement THR-109, Apr. 2015.
- See also: Related Info — http://www.vcu.edu/pcos

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 55 subjects were enrolled, however some subjects failed to meet eligibility criteria resulting in 26 subjects initiating and completing all study phases.
Period: Overall Study
Arm/Group | Metformin
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Metformin
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.9 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 35.0 (7.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders/Non-responders for Each STK11 rs8111699 Genotype (C/G, C/C, G/G)
Description: Responders were defined as those that had a doubling of baseline ovulation rate estimated by self-report of menstrual history.
Time Frame: 9 months
Measure: Number; unit: participants
Groups:
- G/G Genotype; C/G Genotype; C/C Genotype: Metformin tablet, 500 mg per tablet, 2 tablets every 12 hours
Arm/Group | G/G Genotype | C/G Genotype | C/C Genotype
Number analyzed (Participants) | 26 | 26 | 26
participants
  responders | 6 | 7 | 5
  non-responders | 3 | 4 | 1

2. Primary Outcome: Ovulation Rate Over Study Duration for STK11 Genotypes CC, CG and GG
Description: Ovulations were determined by measurement of daily urine pregnanediol-3-glucuronide or weekly progesterone levels over 6-9 months of study duration for each participant. The ovulation rate was calculated as the number of confirmed ovulation events per months of study participation.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: ovulations/month
Arm/Group | G/G Genotype | C/G Genotype | C/C Genotype
Number analyzed (Participants) | 9 | 11 | 6
ovulations/month | 0.47 (0.310) | 0.36 (0.396) | 0.34 (0.336)

3. Secondary Outcome: Determine in Which Genotype(s) Frequency of Ovulation Correlates With Improvement in Reduction in Total Testosterone and Insulin Sensitivity as Measured by the Matsuda Index.
Description: Bivariate fit (RSquare with P values) of ovulation rate post treatment by change in total testosterone and Matsuda Index for each of the 3 genotypes (G/G, C/G, C/C)
Time Frame: 9 months
Population: Individuals that were lost to follow up had missing data on testosterone and OGTT (oral glucose tolerance testing) for Matsuda index.
Measure: Number; unit: Correlation coefficient (r^2)
Arm/Group | G/G Genotype | C/G Genotype | C/C Genotype
Number analyzed (Participants) | 9 | 7 | 3
Correlation coefficient (r^2)
  Ovulation rate vs Testosterone post treatment | 0.138956 | 0.035449 | 0.049263
  Ovulation rate vs Matsuda Index post treatment | 0.27144 | 0.01918 | 0.132059
Statistical Analysis 1: Comparison: G/G Genotype; Test type: Superiority or Other; p = 0.0234, Regression, Linear — Ovulation rate vs Testosterone post-treatment, threshold for statistical significance = p<0.05
Statistical Analysis 2: Comparison: C/G Genotype; Test type: Superiority or Other; p = 0.0740, Regression, Linear — Ovulation rate vs Testosterone post-treatment, threshold for statistical significance = p<0.05
Statistical Analysis 3: Comparison: C/C Genotype; Test type: Superiority or Other; p = 0.4698, Regression, Linear — Ovulation rate vs Testosterone post-treatment, threshold for statistical significance = p<0.05
Statistical Analysis 4: Comparison: G/G Genotype; Test type: Superiority or Other; p = 0.1180, Regression, Linear — Ovulation rate vs Matsuda Index post-treatment, threshold for statistical significance = p < 0.05
Statistical Analysis 5: Comparison: C/G Genotype; Test type: Superiority or Other; p = 0.0311, Regression, Linear — Ovulation rate vs Matsuda Index post-treatment, threshold for statistical significance = p < 0.05
Statistical Analysis 6: Comparison: C/C Genotype; Test type: Superiority or Other; p = 0.1586, Regression, Linear — Ovulation rate vs Matsuda Index post-treatment, threshold for statistical significance = p < 0.05

ADVERSE EVENTS:
Time Frame: For entire 9 months of study plus 30 days after study completion
Arm/Group | Metformin
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 1/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=26)
Anemia (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Interpretations of our findings are limited by our small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No